CLINICAL TRIAL: NCT05359549
Title: Dental Implant Treatment for Two Adjacent Teeth in the Maxillary Aesthetic Region: an Evaluation After 10 Years
Acronym: 2implants
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 202200150
Record Dates: First submitted 2022-03-29; First posted 2022-05-04 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2023-10

CONDITIONS: Missing Teeth
Keywords: dental implants
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Two adjacent dental implants: 25 patients with two missing adjacent teeth in the maxillary aesthetic region which was treated 10 years ago with dental implant placement and an implant-supported restorations.
  Interventions: Device: Two endosseous dental implants (NobelReplace Groovy®) were placed 10 years ago

INTERVENTIONS:
Device: Two endosseous dental implants (NobelReplace Groovy®) were placed 10 years ago — All patients were 10 years ago referred to the Department of Oral and Maxillofacial Surgery (University of Groningen, University Medical Hospital) because of having two failing teeth in the maxillary aesthetic region and were treated with dental implant placement and implant-supported restorations. Patients will have a regular routine control visit (as part of regular follow-up of these patients)

SUMMARY:
* Background Replacement of two missing adjacent teeth is considered a difficult treatment in implant dentistry and even more challenging if located in the anterior region due to aesthetic demands. As well peri-implant bone contour as soft tissue volume is compromised at start of the treatment and difficult to restore. The question is if this reconstruction will be stable in the longterm. Full-scale evaluation of adjacent implant placement with crown rehabilitation in the aesthetic region with a follow-up of at least 10 years is underreported in this field of implant dentistry.
* Main research question The aim of this observational study was to analyze peri-implant bone changes, mucosa levels, aesthetic ratings and patient-reported satisfaction with the maxillary aesthetic region following implant placement with crown restoration after a 10-years follow-up period.
* Design (including population, confounders/outcomes) The study design is an observational study of a group of patients with two missing adjacent teeth in the maxillary aesthetic region which was treated 10 years ago with dental implant placement and an implant-supported restorations.

Outcomes: primary outcome is the change in marginal peri-implant bone level 10 years after placing the definitive restoration. Secondary outcome measures will be implant and restoration survival and changes in interproximal peri-implant mucosa, midfacial peri-implant mucosal level , aesthetic outcome assessed by means of an objective index and patients' satisfaction using a questionnaire.

• Expected results Stable peri-implant bone levels, stable peri-implant soft tissue levels, high implant and restoration survival rate and satisfied patients.

DETAILED DESCRIPTION:
The study design is an observational study of a group of 25 patients with two missing adjacent teeth in the maxillary aesthetic region which was treated 10 years ago with dental implant placement and an implant-supported restorations.

* Inclusion criteria:
* Patients, having two missing teeth in the maxillary aesthetic region, referred to the department of Oral and Maxillofacial Surgery 10 years ago and treated with dental implant placement and implant-supported restorations. At the time of treatment:
* The patient was 18 years or older;
* The failing teeth were an incisor (central or lateral), cuspid or first bicuspid in the maxilla; the adjacent teeth are natural teeth;
* Sufficient healthy and vital bone to insert a dental implant with a minimum length of 10 mm and at least 3.5 mm in diameter with initial stability > 45 Ncm
* The implant site was free from infection;
* Adequate oral hygiene (modified plaque index and modified sulcus bleeding index ≤ 1);
* Sufficient mesio-distal, bucco-lingual, and interocclusal space for placement of an anatomic restoration;
* The patient was capable of understanding and giving informed consent.
* Exclusion criteria at the time of treatment:
* Medical and general contraindications for the surgical procedures;
* Presence of an active and uncontrolled periodontal disease;
* Bruxism;
* Smoking
* A history of local radiotherapy to the head and neck region. All patients were 10 years ago referred to the Department of Oral and Maxillofacial Surgery (University of Groningen, University Medical Hospital) because of having two failing teeth in the maxillary aesthetic region and were treated with dental implant placement and implant-supported restorations. Patients will have a regular routine control visit (as part of regular follow-up of these patients). All data to be collected are part of the routine visit and collected regularly at earlier routine visits, except for the questionnaire. The questionnaire contains a limited number of questions with respect to satisfaction with the aesthetic result. If patients are willing to participate (to use their research data and to fill in the questionnaire), they will be asked to give informed consent by signing a form. After signing, they will be included in the 10-years evaluation as participant. The forms will be collected in the CRF and in the medical record it will be noted that patient has signed the informed consent. Data will be collected during the routine control visit; patients will not have an extra visit for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Patients, having two missing teeth in the maxillary aesthetic region, referred to the department of Oral and Maxillofacial Surgery 10 years ago and treated with dental implant placement and implant-supported restorations. At the time of treatment:

  * The patient was 18 years or older;
  * The failing teeth were an incisor (central or lateral), cuspid or first bicuspid in the maxilla; the adjacent teeth are natural teeth;
  * Sufficient healthy and vital bone to insert a dental implant with a minimum length of 10 mm and at least 3.5 mm in diameter with initial stability > 45 Ncm
  * The implant site was free from infection;
  * Adequate oral hygiene (modified plaque index and modified sulcus bleeding index ≤ 1);
  * Sufficient mesio-distal, bucco-lingual, and interocclusal space for placement of an anatomic restoration;
  * The patient was capable of understanding and giving informed consent.

Exclusion Criteria:

* • Medical and general contraindications for the surgical procedures;

  * Presence of an active and uncontrolled periodontal disease;
  * Bruxism;
  * Smoking
  * A history of local radiotherapy to the head and neck region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients were 10 years ago referred to the Department of Oral and Maxillofacial Surgery (University of Groningen, University Medical Hospital) because of having two failing teeth in the maxillary aesthetic region and were treated with dental implant placement and implant-supported restorations.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Change in peri-implant marginal bone level | Comparison initial radiograph with radiograph after 10 years
  Change in peri-implant marginal bone level along the implant side measured on radiographs in millimetres

SECONDARY OUTCOMES:
Implant survival | 10 years
  Percentage of initially placed of dental implants present after 10 years
Restoration survival | 10 years
  Survival of implant restorations after 10 years
Peri-implant soft tissue health | Status at 10 years
  Health of peri-implant soft tissues after 10 years measured with an ordinal index
Patient satisfaction | Satisfaction at 10 years
  Satisfaction of patients measured with an VAS scale in questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Henny JA Meijer, Prof, Principal Investigator — University Medical Center Groningen
Locations (1):
- Dept Oral and Maxillofacial Surgery UMCG, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request

REFERENCES:
- [Background] Tymstra N, Raghoebar GM, Vissink A, Den Hartog L, Stellingsma K, Meijer HJ. Treatment outcome of two adjacent implant crowns with different implant platform designs in the aesthetic zone: a 1-year randomized clinical trial. J Clin Periodontol. 2011 Jan;38(1):74-85. doi: 10.1111/j.1600-051X.2010.01638.x. Epub 2010 Nov 10. PMID 21062337
- [Background] Van Nimwegen WG, Raghoebar GM, Stellingsma K, Tymstra N, Vissink A, Meijer HJ. Treatment Outcome of Two Adjacent Implant-Supported Restorations with Different Implant Platform Designs in the Esthetic Region: A Five-Year Randomized Clinical Trial. Int J Prosthodont. 2015 Sep-Oct;28(5):490-8. doi: 10.11607/ijp.4199. PMID 26340009